CLINICAL TRIAL: NCT00135668
Title: A Phase 2 Multicenter, Randomized, Double-blind, Parallel Group, Dose-ranging, Effect-controlled Study to Determine the Pharmacokinetics and Pharmacodynamics of Sodium Nitroprusside in Pediatric Subjects
Brief Title: Dose-response Study of Sodium Nitroprusside in Children Requiring Controlled Hypotension in the Operating Room
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: Stanford University (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-2003-09-DR; N01HD43386-7-0-1 (NIH)
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Hypotension
Keywords: children; sodium nitroprusside; controlled hypotension; dose-response; pharmacokinetics; pharmacodynamics; safety; efficacy
MeSH Terms: conditions — Hypotension | interventions — Nitroprusside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.3 mcg/kg/min (Active Comparator): Infusion of Sodium Nitroprusside began only after a 5-minute period of stable anesthesia or sedation (no changes in dosages). The infusion rate during the blinded study drug period was increased in a step-wise fashion to the full dose rate as follows: 5 ± 1 minutes at 1/3 of the full rate; 5 ± 1 minutes at 2/3 of the full rate; and 20 minutes at the full dose rate (ie, 30 minutes total). The full infusion rate was 0.6 mL/kg/hr; 2/3 of the full rate was 0.4 mL/kg/hr; and 1/3 of the full rate was 0.2 mL/kg/hr. After titration to the full dose of blinded study drug, blinded infusion dosage adjustments were not permitted during the blinded study drug administration period. The blinded infusion dosage continued for the 30 minutes unless clinical events demanded a change for safety reasons.
  Interventions: Drug: Nitroprusside
- 1 mcg/kg/min (Active Comparator): Infusion of Sodium Nitroprusside began only after a 5-minute period of stable anesthesia or sedation (no changes in dosages). The infusion rate during the blinded study drug period was increased in a step-wise fashion to the full dose rate as follows: 5 ± 1 minutes at 1/3 of the full rate; 5 ± 1 minutes at 2/3 of the full rate; and 20 minutes at the full dose rate (ie, 30 minutes total). The full infusion rate was 0.6 mL/kg/hr; 2/3 of the full rate was 0.4 mL/kg/hr; and 1/3 of the full rate was 0.2 mL/kg/hr. After titration to the full dose of blinded study drug, blinded infusion dosage adjustments were not permitted during the blinded study drug administration period. The blinded infusion dosage continued for the 30 minutes unless clinical events demanded a change for safety reasons.
  Interventions: Drug: Nitroprusside
- 2 mcg/kg/min (Active Comparator): Infusion of Sodium Nitroprusside began only after a 5-minute period of stable anesthesia or sedation (no changes in dosages). The infusion rate during the blinded study drug period was increased in a step-wise fashion to the full dose rate as follows: 5 ± 1 minutes at 1/3 of the full rate; 5 ± 1 minutes at 2/3 of the full rate; and 20 minutes at the full dose rate (ie, 30 minutes total). The full infusion rate was 0.6 mL/kg/hr; 2/3 of the full rate was 0.4 mL/kg/hr; and 1/3 of the full rate was 0.2 mL/kg/hr. After titration to the full dose of blinded study drug, blinded infusion dosage adjustments were not permitted during the blinded study drug administration period. The blinded infusion dosage continued for the 30 minutes unless clinical events demanded a change for safety reasons
  Interventions: Drug: Nitroprusside
- 3 mcg/kg/min (Active Comparator): Infusion of Sodium Nitroprusside began only after a 5-minute period of stable anesthesia or sedation (no changes in dosages). The infusion rate during the blinded study drug period was increased in a step-wise fashion to the full dose rate as follows: 5 ± 1 minutes at 1/3 of the full rate; 5 ± 1 minutes at 2/3 of the full rate; and 20 minutes at the full dose rate (ie, 30 minutes total). The full infusion rate was 0.6 mL/kg/hr; 2/3 of the full rate was 0.4 mL/kg/hr; and 1/3 of the full rate was 0.2 mL/kg/hr. After titration to the full dose of blinded study drug, blinded infusion dosage adjustments were not permitted during the blinded study drug administration period. The blinded infusion dosage continued for the 30 minutes unless clinical events demanded a change for safety reasons
  Interventions: Drug: Nitroprusside

INTERVENTIONS:
Drug: Nitroprusside — Study drug was infused via a dedicated peripheral intravenous catheter or via a dedicated lumen of a multi-orifice central venous catheter. Infusion pumps capable of reliable delivery at low infusion rates (to 0.1 mL/hr) were used.Study drug was dispensed to the sites in 2 mL vials containing 25 mg/mL of sodium nitroprusside. The pharmacist prepared and dispensed the study drug, and supplied blinded study drug for each subject according to a randomization assignment generated by the IVRS (Interactive Voice Response System).
  Other Names: Sodium Nitroprusside IV infusion 0.3 mcg/kg/ min
  Arms: 0.3 mcg/kg/min
Drug: Nitroprusside — Study drug was infused via a dedicated peripheral intravenous catheter or via a dedicated lumen of a multi-orifice central venous catheter. Infusion pumps capable of reliable delivery at low infusion rates (to 0.1 mL/hr) were used.Study drug was dispensed to the sites in 2 mL vials containing 25 mg/mL of sodium nitroprusside. The pharmacist prepared and dispensed the study drug, and supplied blinded study drug for each subject according to a randomization assignment generated by the IVRS.
  Other Names: Sodium Nitroprusside IV infusion 1 mcg/kg/ min
  Arms: 1 mcg/kg/min
Drug: Nitroprusside — Study drug was infused via a dedicated peripheral intravenous catheter or via a dedicated lumen of a multi-orifice central venous catheter. Infusion pumps capable of reliable delivery at low infusion rates (to 0.1 mL/hr) were used.Study drug was dispensed to the sites in 2 mL vials containing 25 mg/mL of sodium nitroprusside. The pharmacist prepared and dispensed the study drug, and supplied blinded study drug for each subject according to a randomization assignment generated by the IVRS.
  Other Names: Sodium Nitroprusside IV infusion 2 mcg/kg/ min
  Arms: 2 mcg/kg/min
Drug: Nitroprusside — Study drug was infused via a dedicated peripheral intravenous catheter or via a dedicated lumen of a multi-orifice central venous catheter. Infusion pumps capable of reliable delivery at low infusion rates (to 0.1 mL/hr) were used.Study drug was dispensed to the sites in 2 mL vials containing 25 mg/mL of sodium nitroprusside. The pharmacist prepared and dispensed the study drug, and supplied blinded study drug for each subject according to a randomization assignment generated by the IVRS
  Other Names: Sodium Nitroprusside IV infusion 3 mcg/kg/ min
  Arms: 3 mcg/kg/min

SUMMARY:
Sodium nitroprusside (SNP) has been approved for control of blood pressure in adults, yet there are no controlled studies in children. The purpose of this study is to determine the efficacy and safety of sodium nitroprusside in children who will be having surgery, and who require blood pressure lowering in order to decrease the amount of blood loss during their surgery.

DETAILED DESCRIPTION:
The trial is a multicenter randomized, double-blind, parallel group, dose-ranging, effect-controlled study examining the effects of sodium nitroprusside in pediatric subjects requiring relative hypotension during a surgical or medical procedure. The goal is to establish the starting and maximum infusion rates that afford optimum blood pressure control in children and a safe dosing regimen in children. The objective is to describe the relationship between the infusion rate of nitroprusside and changes in blood pressure.

The specific aims of this trial are:

1. To define the onset and offset of blood pressure lowering effects of nitroprusside to obtain adequate instructions for dose titration in the pediatric population.
2. To construct a dose-response model that defines the relationship between nitroprusside infusion rate and changes in blood pressure in pediatric subjects.
3. To assess the safety of nitroprusside administration in pediatric subjects requiring controlled reduction of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

Study subjects must meet all of the following criteria:

* Subject is less than 17 years of age
* Neonates must be full-term gestation and have a body weight of at least 2.5 kg
* Subject requires pharmacologically-induced hypotension for acute blood pressure management for surgery or other invasive procedure, e.g., cerebral artery embolization
* Duration of the subject's controlled hypotension is expected to be ≥ 2 hours
* Subject requires general anesthesia with endotracheal intubation
* Subject requires placement of intra-arterial line during the surgical or medical procedure
* The subject's parent or legal guardian gives permission (informed consent) and subject gives assent when appropriate.

Exclusion Criteria:

Subjects will be excluded if any of the following criteria exist:

* Subject has a known allergy to SNP
* Subject has a known mitochondrial cytopathy with a disorder of oxidative phosphorylation or of respiratory chain enzymes
* Subject has a contraindication to vasodilator therapy for control of blood pressure during surgery or procedures
* Subject has participated in other clinical trials for investigational drugs and/or devices within 30 days prior to enrollment
* Subject has any serious medical condition which, in the opinion of the investigator, is likely to interfere with study procedures
* Subject is moribund (death likely to occur within 48 hours)
* Subject has a positive result for the urine or serum human chorionic gonadotropin (HCG) test administered at screening.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hammer, MD, Principal Investigator — Stanford University; Scott Schulman, MD, Principal Investigator — Duke University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Drover DR, Hammer GB, Barrett JS, Cohane CA, Reece T, Zajicek A, Schulman SR. Evaluation of sodium nitroprusside for controlled hypotension in children during surgery. Front Pharmacol. 2015 Jul 6;6:136. doi: 10.3389/fphar.2015.00136. eCollection 2015. PMID 26217225
- [Derived] Hammer GB, Connolly SG, Schulman SR, Lewandowski A, Cohane C, Reece TL, Anand R, Mitchell J, Drover DR. Sodium nitroprusside is not associated with metabolic acidosis during intraoperative infusion in children. BMC Anesthesiol. 2013 Apr 30;13:9. doi: 10.1186/1471-2253-13-9. PMID 23631460

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 206 participants were randomized to be dosed with one of 4 differed SNP infusion rates.
Pre-assignment Details: Of the 206 randomized participants, 3 discontinued pre-operatively and 203 participants completed the study and no patients discontinued the study post operative. Participants counted as completing the study may have stopped the blinded study drug period early but continued on to the open-label study drug period and follow-up period.
Groups:
- 0.3 μg/kg/Min: Rate of SNP infusion during blinded study drug period
  Patients who were randomized and never received a dose of study drug did not contribute data to any analysis population. The following three analysis populations were included in the study:
  Intent-to-Treat Safety (ITT S) Population consisted of all consented and randomized patients who received any amount of study drug
  Intent-to-Treat Efficacy Evaluable (ITT E) Population consisted of randomized and treated patients who had a pre treatment Baseline MAP and a second MAP determined within 30 minutes of study drug infusion at the starting dose
  Intent-to-Treat Completer (ITT C) Population consisted of all randomized and treated patients who completed the 30-minute blinded study drug period. The ITT C population is indicated by the participants who completed 'period 2.
  P
- 1 μg/kg/Min: Rate of SNP infusion during blinded study drug period
  Patients who were randomized and never received a dose of study drug did not contribute data to any analysis population. The following three analysis populations were included in the study:
  Intent-to-Treat Safety (ITT S) Population consisted of all consented and randomized patients who received any amount of study drug
  Intent-to-Treat Efficacy Evaluable (ITT E) Population consisted of randomized and treated patients who had a pre treatment Baseline MAP and a second MAP determined within 30 minutes of study drug infusion at the starting dose
  Intent-to-Treat Completer (ITT C) Population consisted of all randomized and treated patients who completed the 30-minute blinded study drug period. The ITT C population is indicated by the participants who completed 'period 2.
  .
- 2 μg/kg/Min; 3 μg/kg/Min: Rate of SNP infusion during blinded study drug period
  Patients who were randomized and never received a dose of study drug did not contribute data to any analysis population. The following three analysis populations were included in the study:
  Intent-to-Treat Safety (ITT S) Population consisted of all consented and randomized patients who received any amount of study drug
  Intent-to-Treat Efficacy Evaluable (ITT E) Population consisted of randomized and treated patients who had a pre treatment Baseline MAP and a second MAP determined within 30 minutes of study drug infusion at the starting dose
  Intent-to-Treat Completer (ITT C) Population consisted of all randomized and treated patients who completed the 30-minute blinded study drug period. The ITT C population is indicated by the participants who completed 'period 2.
Period: Overall Study - Randomized to be Dosed
Arm/Group | 0.3 μg/kg/Min | 1 μg/kg/Min | 2 μg/kg/Min | 3 μg/kg/Min
Started | 51 | 49 | 55 | 51
Completed | 50 | 49 | 53 | 51
Not Completed | 1 | 0 | 2 | 0
Not completed — Discontinued pre-operatively | 1 | 0 | 2 | 0
Period: Blinded Treatment Phase-Randomized/Dosed
Arm/Group | 0.3 μg/kg/Min | 1 μg/kg/Min | 2 μg/kg/Min | 3 μg/kg/Min
Started | 50 | 49 | 53 | 51
Completed | 38 | 23 | 13 | 18
Not Completed | 12 | 26 | 40 | 33

BASELINE CHARACTERISTICS:
Population: 211 participants were enrolled in the study; 206 were randomized, 5 discontinued preoperatively.
  Of the 206, 3 discontinued preoperatively after randomization resulting in 203 participants who completed the study. These 203 participants constituted the baseline population.
Groups:
- 0.3 mcg/kg/Min: Infusion rate scheduled to be titrated during the blinded phase to 0.3 mcg/kg/min
- 1 mcg/kg/Min: Infusion rate scheduled to be titrated during the blinded phase to 1 mcg/kg/min
- 2 mcg/kg/Min: Infusion rate scheduled to be titrated during the blinded phase to 2 mcg/kg/min
- 3 mcg/kg/Min: Infusion rate scheduled to be titrated during the blinded phase to 3 mcg/kg/min
- Total: Total of all reporting groups
Arm/Group | 0.3 mcg/kg/Min | 1 mcg/kg/Min | 2 mcg/kg/Min | 3 mcg/kg/Min | Total
Number analyzed (Participants) | 50 | 49 | 53 | 51 | 203
Age, Customized [Mean (Standard Deviation); unit: Months] | 110.30 (75.424) | 114.74 (71.479) | 114.21 (73.864) | 111.30 (76.429) | 112.64 (73.610)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 20 | 19 | 74
  Male | 36 | 28 | 33 | 32 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 12 | 13 | 47
  Not Hispanic or Latino | 39 | 38 | 41 | 38 | 156
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Arterial Pressure (MAP) From the Baseline MAP
Description: From the Baseline MAP until the end of the blinded phase; scheduled for 30 min
Time Frame: Approximately 30 minutes
Population: Change from Baseline in MAP across the Sodium Nitroprusside (SNP) dose groups by mean at Baseline, 30 mins (LOCF), and change from Baseline for the ITT Efficacy Evaluable Population consisted of randomized and treated patients who had a pre-treatment Baseline MAP and a second MAP determined within 30 mins of study drug infusion at the starting dose
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- 0.3 mcg/kg/Min; 1 mcg/kg/Min; 2 mcg/kg/Min; 3 mcg/kg/Min: Rate of SNP infusion during blinded study drug period
- Total: Total result
Arm/Group | 0.3 mcg/kg/Min | 1 mcg/kg/Min | 2 mcg/kg/Min | 3 mcg/kg/Min | Total
Number analyzed (Participants) | 50 | 49 | 53 | 51 | 203
mm Hg
  Baseline Observed | 76.3 (11.37) | 76.9 (14.5) | 73.5 (11.5) | 76.3 (12.06) | 75.7 (12.37)
  30 Minutes LOCF(last observation carried forward) | 65.3 (13.30) | 59.9 (15.43) | 53.5 (12.09) | 59.6 (17.82) | 59.5 (15.28)
  Change from Baseline | -11.0 (15.68) | -17.0 (12.88) | -20.0 (15.95) | -16.6 (18.63) | -16.2 (16.16)
Statistical Analysis 1: Comparison: Total; Paired t-test used to test the null hypothesis of no change in MAP from baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired t-test used; Mean Difference (Final Values) = -16.2, 95% CI 2-sided [-18.44 to -13.97], Standard Deviation 16.16
Statistical Analysis 2: Comparison: 0.3 mcg/kg/Min; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -11.0, 95% CI 2-sided [-15.45 to -6.55], Standard Deviation 15.68
Statistical Analysis 3: Comparison: 1 mcg/kg/Min; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -17.0, 95% CI 2-sided [-20.70 to -13.30], Standard Deviation 12.88
Statistical Analysis 4: Comparison: 2 mcg/kg/Min; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -20.0, 95% CI 2-sided [-24.38 to -15.58], Standard Deviation 15.95
Statistical Analysis 5: Comparison: 3 mcg/kg/Min; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -16.6, 95% CI 2-sided [-21.87 to -11.39], Standard Deviation 18.63

2. Primary Outcome: Overall Summary of Tolerability/Adverse Events (AEs) for ITT Safety Population
Description: Treatment-emergent AEs (TEAEs) were defined as an AE experienced by the patient that was either first observed after the initiation of study drug (blinded or open-label) or represented an exacerbation (usually in severity) of a pre existing condition observed prior to treatment. Subjects will be followed for 30 days after discontinuation of study drug. The occurrence of Serious Adverse Events (SAEs) will be monitored for 30 days.
Time Frame: 30 days
Population: ITT Safety Population consisted of all consented and randomized patients who received any amount of study medication
Measure: Number; unit: participants
Groups:
- 0.3 mcg/kg/Min; 1 mcg/kg/Min; 2 mcg/kg/Min; 3 mcg/kg/Min: Rate of SNP Infusion
- Total: Overall
Arm/Group | 0.3 mcg/kg/Min | 1 mcg/kg/Min | 2 mcg/kg/Min | 3 mcg/kg/Min | Total
Number analyzed (Participants) | 50 | 49 | 53 | 51 | 203
participants
  N of participants with at least one TEAE | 50 | 49 | 53 | 51 | 203
  N of participants with at least one TESAE | 5 | 4 | 5 | 4 | 18
  N with TEAE leading to study drug withdrawal | 19 | 18 | 13 | 16 | 66
  N of participants with MILD TEAE | 8 | 10 | 7 | 8 | 33
  N of participants with MODERATE TEAE | 19 | 19 | 20 | 15 | 73
  N of participants with SEVERE TEAE | 23 | 20 | 26 | 28 | 97
  N of participants with probably related TEAE | 29 | 32 | 40 | 36 | 137
  N of participants with possibly related TEAE | 12 | 6 | 2 | 9 | 29
  N of participants with Probably NOT related TEAE | 1 | 5 | 0 | 3 | 9
  N of participants with NOT related TEAE | 8 | 6 | 11 | 3 | 28
  N of Deaths | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline MAP Nitroprusside Infusion During the Blinded Infusion;
Description: Change From Baseline in MAP (mmHg) After 20 and 25 Minutes Double-Blind Infusion (Overall) for ITT Efficacy Evaluable Population.
Time Frame: 25 minutes
Population: ITT Efficacy Evaluable Population consisted of randomized and treated patients who had a pre-treatment Baseline MAP and a second MAP determined within 25 minutes of study drug infusion at the starting dose.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- 0.3 mcg/kg/Min: N for 20 min observation - 42 N for 25 min observation - 39
- 1 mcg/kg/Min: N for 20 min observation - 27 N for 25 min observation - 24
- 2 mcg/kg/Min: N for 20 min observation - 19 N for 25 min observation - 15
- 3 mcg/kg/Min: N for 20 min observation - 26 N for 25 min observation - 20
- Total: N for 20 min observation - 114 N for 25 min observation - 98
Arm/Group | 0.3 mcg/kg/Min | 1 mcg/kg/Min | 2 mcg/kg/Min | 3 mcg/kg/Min | Total
Number analyzed (Participants) | 50 | 49 | 53 | 51 | 203
mm Hg
  Baseline (BL) Observed (n = 50,49,53,51,203) | 76.3 (11.37) | 76.9 (14.50) | 73.5 (11.50) | 76.3 (12.06) | 75.7 (12.37)
  20 Mins Observed (n = 42,27,19,26,114): number analyzed (Participants) | 42 | 27 | 19 | 26 | 114
  20 Mins Observed (n = 42,27,19,26,114) | 69.6 (11.29) | 73.2 (15.97) | 62.3 (13.58) | 65.8 (12.73) | 68.4 (13.57)
  Change from BL - 20 mins (n = 42,27,19,26,114): number analyzed (Participants) | 42 | 27 | 19 | 26 | 114
  Change from BL - 20 mins (n = 42,27,19,26,114) | -7.5 (14.38) | -10.0 (16.37) | -11.1 (16.42) | -12.5 (14.09) | -9.8 (15.08)
  25 mins observed (n = 39,24,15,20,98): number analyzed (Participants) | 39 | 24 | 15 | 20 | 98
  25 mins observed (n = 39,24,15,20,98) | 69.5 (12.15) | 64.4 (10.30) | 60.5 (10.53) | 66.4 (13.07) | 66.2 (11.94)
  Change from BL - 25 mins (n = 39,24,15,20,98): number analyzed (Participants) | 39 | 24 | 15 | 20 | 98
  Change from BL - 25 mins (n = 39,24,15,20,98) | -6.9 (11.80) | -18.2 (14.69) | -10.2 (13.82) | -11.7 (16.16) | -11.1 (14.21)

4. Secondary Outcome: Infusion Rate of Sodium Nitroprusside That Reduces MAP to a Predetermined Clinically Meaningful Target Value +/- 10%;
Description: Infusion rate of sodium nitroprusside at which a predetermined clinically meaningful target value (+/- 10%) of MAP was achieved during study drug administration
Time Frame: Up to the end of open label treatment (Approximately 120 minutes)
Population: The Analysis population included the participants in the ITT Efficacy evaluable population who achieved target MAP. ITT Efficacy Evaluable Population consisted of randomized and treated patients who had a pre-treatment Baseline MAP and a second MAP determined within 30 minutes of study drug.
Measure: Mean (Standard Deviation); unit: mcg/kg/min
Arm/Group | 0.3 mcg/kg/Min | 1 mcg/kg/Min | 2 mcg/kg/Min | 3 mcg/kg/Min | Total
Number analyzed (Participants) | 48 | 49 | 52 | 51 | 200
mcg/kg/min | 0.47 (0.519) | 0.70 (0.346) | 1.21 (0.678) | 1.86 (0.922) | 1.07 (0.843)

5. Secondary Outcome: Number of Participants Who Reach Target MAP;
Description: Blinded Study Drug Administration Period: Started with study drug administration following stabilization of anesthesia. Patients were administered a blinded dose of SNP for up to 30 mins.
  This period ended at the start of open-label study drug infusion or at the completion of the blinded infusion if no open-label study drug was given. The follow-up period immediately followed for those patients not receiving open-label infusion.
  Blinded Treatment Phase II - gap between the end of blinded study drug infusion and the start of open-label study drug infusion
  Open-label treatment phase began with the start of open-label study drug infusion and was at least 90 mins in duration. SNP was initiated at a dose deemed appropriate by the investigator and was gradually adjusted to reach a target MAP based on clinical presentation and needs of the patient. Target MAP was not to be < 50 mmHg (40 mmHg for patients < 30 days of age). This period ended at the completion of open-label infusion.
Time Frame: To the end of open label treatment (approximately 120 minutes)
Population: ITT Efficacy Evaluable Population consisted of randomized and treated patients who had a pre-treatment Baseline MAP and a second MAP determined within 30 minutes of study drug
Measure: Number; unit: participants
Groups:
- 0.3 mcg/kg/Min: Infusion rate scheduled to be titrated to 0.3 mcg/kg/min
- 1 mcg/kg/Min: Infusion rate scheduled to be titrated to 1 mcg/kg/min
- 2 mcg/kg/Min: Infusion rate scheduled to be titrated to 2 mcg/kg/min
- 3 mcg/kg/Min: Infusion rate scheduled to be titrated to 3 mcg/kg/min
Arm/Group | 0.3 mcg/kg/Min | 1 mcg/kg/Min | 2 mcg/kg/Min | 3 mcg/kg/Min | Total
Number analyzed (Participants) | 50 | 49 | 53 | 51 | 203
participants
  Achieved target MAP | 48 | 49 | 52 | 51 | 200
  Did NOT achieve target MAP | 2 | 0 | 0 | 0 | 2
  Not determined | 0 | 0 | 1 | 0 | 1
  Achieved during the blinded treatment | 35 | 36 | 38 | 39 | 148
  Achieved during Blinded Phase II | 0 | 4 | 8 | 7 | 19
  Achieved during Open-label Treatment | 13 | 9 | 6 | 5 | 33

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the first 4 stages stages (prestudy drug administration, Blinded period, Open period,Follow-up period) of the study totalling upto 16 days.Serious adverse events was monitored for additional 30 days after follow-up
Description: Treatment-emergent AEs (TEAEs) were defined as an AE experienced by the patient that was either first observed after the initiation of study drug (blinded or open-label) or represented an exacerbation (usually in severity) of a pre existing condition observed prior to treatment.Serious Adverse events include AEs leading to study drug withdrawal
Groups:
- 0.3 μg/kg/Min; 1 μg/kg/Min; 2 μg/kg/Min: Rate of SNP infusion during blinded study drug period
- 3 μg/kg/Min: Rate of study drug infusion during blinded study drug period
Arm/Group | 0.3 μg/kg/Min | 1 μg/kg/Min | 2 μg/kg/Min | 3 μg/kg/Min
Serious Adverse Events (participants affected / at risk) | 24/50 | 22/49 | 18/53 | 20/51
Other Adverse Events (participants affected / at risk) | 50/50 | 49/49 | 53/53 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3 μg/kg/Min (N=50) | 1 μg/kg/Min (N=49) | 2 μg/kg/Min (N=53) | 3 μg/kg/Min (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Pseudocyst (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Postoperative Infection (Infections and infestations) | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Serratia Infection (Infections and infestations) | 1 | 0 | 0 | 0
Cerebrospinal fluid Leakage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion site extravasation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Operative Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood Pressure decreased (Investigations) | 1 | 2 | 1 | 1
Cardiac output decreased (Investigations) | 1 | 0 | 0 | 0
Central Venous pressure increased (Investigations) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Cauda Equina Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Hypotonic Urinary Bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Rebound Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 16 | 15 | 11 | 15
Superior mesenteric artery syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Heart Rate increased (Investigations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 μg/kg/Min (N=50) | 1 μg/kg/Min (N=49) | 2 μg/kg/Min (N=53) | 3 μg/kg/Min (N=51)
Anaemia (Blood and lymphatic system disorders) | 17 (17) | 13 (13) | 8 (8) | 11 (11)
Coagulopathy (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 4 (4) | 5 (5)
Tachycardia (Cardiac disorders) | 6 (6) | 11 (11) | 8 (8) | 6 (6)
Eye Swelling (Eye disorders) | 4 (4) | 4 (4) | 4 (4) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (6) | 7 (7) | 7 (7) | 6 (6)
Vomiting (Gastrointestinal disorders) | 14 (14) | 13 (13) | 21 (21) | 16 (16)
Face Oedema (General disorders) | 6 (6) | 4 (4) | 8 (8) | 5 (5)
Pyrexia (General disorders) | 16 (16) | 16 (16) | 15 (15) | 24 (24)
Blood Pressure Increased (Investigations) | 5 (5) | 4 (4) | 3 (3) | 1 (1)
Oxygen saturation decreased (Investigations) | 3 (3) | 3 (3) | 5 (5) | 6 (6)
Urine Output decreased (Investigations) | 8 (8) | 10 (10) | 9 (9) | 12 (12)
Acidosis (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 7 (7) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 3 (3) | 3 (3)
Metabolic Acidosis (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 4 (4) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Periorbital Oedema (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 6 (6) | 5 (5)
Haemorrhage (Vascular disorders) | 6 (6) | 4 (4) | 7 (7) | 2 (2)
Hypertension (Vascular disorders) | 10 (10) | 11 (11) | 12 (12) | 19 (19)
Hypotension (Vascular disorders) | 35 (35) | 37 (37) | 40 (40) | 41 (41)
Rebound Hypertension (Vascular disorders) | 7 (7) | 10 (10) | 15 (15) | 16 (16)
Swelling Face (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 8 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No